CLINICAL TRIAL: NCT03925610
Title: Recovery of Ventilation After General Anesthesia in Morbidly Obese Patients Who Are Treated With Opioids: A Preliminary Investigation
Brief Title: Recovery of Ventilation After General Anesthesia in Morbidly Obese Patients
Status: Terminated | Type: Observational
Why Stopped: Lack of resources and COVID-related closure in 2020.
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Anthony Doufas, Professor, Department of Anesthesiology, Perioperative and Pain Medicine, Stanford University
Other Study IDs: IRB-49407
Record Dates: First submitted 2019-04-21; First posted 2019-04-24 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Morbid Obesity; Opioid-Related Disorders; Surgery--Complications; Sleep Apnea Syndromes
Keywords: Morbid obesity; Opioid-induced ventilatory depression; Bariatric surgery; Sleep apnea
MeSH Terms: conditions — Obesity, Morbid; Opioid-Related Disorders; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Morbidly obese patients with moderate-to-severe OSA: Morbidly obese patients recovering from general anesthesia after weight loss surgery (gastric bypass and sleeve placement) surgery.
  All patients will undergo preoperative and postoperative continuous transcutaneous and intermittent arterial blood PCO2 monitoring.
  Sedation depth and pain assessment will be performed in the post-anesthesia care unit (PACU). Fentanyl only will be administered during surgery and in PACU to provide analgesia (verbal numerical score ≤ 3).
  A total of 9, 10-mL blood samples (including a preoperative blank sample) will be obtained throughout the study period (1 preoperatively, 4 intraoperatively and 4 in the PACU) to measure fentanyl concentration in the plasma. Five 1-mL samples will be used to determine arterial PCO2.
- Morbidly obese patients with no or mild OSA: Morbidly obese patients recovering from general anesthesia after weight loss surgery (gastric bypass and sleeve placement) surgery.
  All patients will undergo preoperative and postoperative continuous transcutaneous and intermittent arterial blood PCO2 monitoring.
  Sedation depth and pain assessment will be performed in the post-anesthesia care unit (PACU). Fentanyl only will be administered during surgery and in PACU to provide analgesia (verbal numerical score ≤ 3).
  A total of 9, 10-mL blood samples (including a preoperative blank sample) will be obtained throughout the study period (1 preoperatively, 4 intraoperatively and 4 in the PACU) to measure fentanyl concentration in the plasma. Five 1-mL samples will be used to determine arterial PCO2.

SUMMARY:
This is an observational study of morbidly obese patients recovering from general anesthesia after weight-loss surgery. The investigators aim to assess ventilatory function and how this is influenced by the diagnosis of obstructive sleep apnea (OSA), baseline ventilatory status, as well as pharyngeal collapsibility of patients who are recovering from anesthesia and treated for pain with opioids. The investigators hypothesize that patients with OSA, chronic (baseline) hypoventilation and increased pharyngeal collapsibility, will be more vulnerable to opioid-induced ventilatory depression.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) increases the risk for pulmonary complications in the first 24 hours after surgery, by more than 3-fold, suggesting an enhanced sensitivity to opioid-induced ventilatory depression (OIVD), in this patient population. Obesity and OSA, two highly comorbid conditions, are common among victims of postoperative life-threatening or fatal OIVD and increased somnolence preceding the onset of a critical event, is an almost ubiquitous clinical finding.

These clinical observations are in agreement with recent evidence that decreased wakefulness is an important contributory mechanism of OIVD in OSA patients who receive opioid analgesia in the postoperative period. Studies that examined the effect of opioids on breathing in awake, sleeping, or anesthetized patients with OSA, support overall that OSA is not associated with increased sensitivity to OIVD in awake subjects. In contrast, diminished wakefulness has been shown to worsen, leave unaffected, or even slightly improve breathing and oxygenation in patients with OSA, who are treated opioids.

Decrease in the tonic activity of the pharyngeal muscles with the progression from wakefulness to sleep, contributes to increased airway resistance and the predisposition to airway occlusion. This effect of sleep on the patency of pharyngeal airway seems to be more pronounced in patients with OSA, who present with increased genioglossus muscle activity during wakefulness taken as evidence for a neural compensation to maintain adequate airflow in the presence of anatomical airway narrowing.

It can thus be suggested that during pharmacological suppression of consciousness, like when recovering from anesthesia, patients with OSA will experience more severe sleep-disordered breathing and consequently be more vulnerable to OIVD, compared to normal subjects.

Specific Aims

Specific Aim 1: To assess opioid-induced ventilatory depression in morbidly obese patients with OSA, who recover from general anesthesia and are treated for pain with fentanyl. We will develop a pharmacodynamic model for OIVD to assess the effect of OSA status (i.e., moderate-to-severe OSA vs. no or mild OSA) on the probability for TcPCO2 to exceed a pre-specified threshold during recovery from anesthesia.

Specific Aim 2: To assess the effect of baseline TcPCO2 on the probability for TcPCO2 to exceed a pre-specified threshold during recovery from anesthesia, independently of the OSA status.

Specific Aim 3: To assess the effect of the minimum positive airway pressure (minPAP) that prevents obstructive breathing during sleep (estimated during in-lab polysomnography) on the probability for TcPCO2 to exceed a pre-specified threshold, during recovery from anesthesia.

Hypotheses:

1. Patients with moderate-to-severe OSA will demonstrate a higher probability for exceeding a pre-specified threshold for TcPCO2, compared to those with mild or no OSA, during recovery from general anesthesia.
2. Patients who present with higher TcPCO2 at baseline, will present with a higher probability to exceed a pre-specified threshold for TcPCO2, independently of their OSA status, compared to those with normal ventilatory control at baseline, during recovery from anesthesia.
3. Patients with higher therapeutic PAP level (hence more collapsible airway) will be more sensitive to fentanyl-induced ventilatory depression and will thus demonstrate a higher probability for exceeding a pre-specified threshold for TcPCO2 during recovery from anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) equal or greater than 35 kg/m2.
* American Society of Anesthesiologists (ASA) physical status I - III patients.
* Scheduled to undergo laparoscopic roux-en-Y gastric bypass or gastric sleeve placement surgery for weight loss.

Exclusion Criteria:

* Chronic obstructive pulmonary disorder (COPD).
* Treatment with continuous positive airway pressure (CPAP) in the past three months.
* Severe neurological, cardiopulmonary, psychiatric, or untreated thyroid disorder.
* Chronic pain condition that was being treated with opioids.
* Patients with a hematocrit lower than 35%.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Morbidly obese patients who are eligible for weight-loss surgery.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Probability for TcPCO2 / PaCO2 to exceed a pre-specified threshold during recovery from anesthesia. | PACU period (approximate duration of about 1.5h).
  Probability for TcPCO2 / PaCO2 to exceed a pre-specified threshold during recovery from anesthesia.

SECONDARY OUTCOMES:
The effect of baseline ventilation on the primary outcome | PACU period (approximate duration of about 1.5h)
  Effect of baseline ventilation, expressed as transcutaneous and arterial PCO2, on the primary outcome.
The effect of the minimum PAP on the primary outcome. | PACU period (approximate duration of 1.5h)
  The effect of the minimum positive airway pressure (minPAP) that prevents obstructive breathing during sleep (estimated during in-lab polysomnography) on the probability for TcPCO2 /PaCO2 to exceed a pre-specified threshold

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Doufas, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No